CLINICAL TRIAL: NCT06429852
Title: Examining the Efficacy, Feasibility, and Acceptability of the DeST-ACT: Trauma-Focused Acceptance and Commitment Therapy Program on Life Satisfaction in Earthquake Survivors
Brief Title: Efficacy, Feasibility, and Acceptability of the DeST-ACT: Trauma-Focused Acceptance and Commitment Therapy Program
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CanSagligi Foundation (Other)
Responsible Party: Principal Investigator, Sevinc Ulusoy, Principal Investigator, CanSagligi Foundation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSV202403
Record Dates: First submitted 2024-05-21; First posted 2024-05-28 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Trauma and Stressor Related Disorders
MeSH Terms: conditions — Trauma and Stressor Related Disorders

STUDY DESIGN:
Intervention Model Description: The study will be a quantitative, randomized controlled trial with two groups, including a pre-test and repeated post-tests.
Masking Description: Randomization will be conducted by a research assistant using an internet-based program following the pre-test. The pre-test and post-tests will be administered by a different researcher who is blinded to the study. The therapy program will be conducted by independent therapists who are also blinded to the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DeST-ACT Intervention Group (Experimental): Participants in the intervention group will undergo the DeST-ACT psychosocial intervention. This program includes a 4-session online intervention supplemented with self-help materials. These materials comprise concise texts designed to reinforce the skills covered in each session.
  Interventions: Behavioral: The DeST-ACT Trauma-Focused Acceptance and Commitment Therapy Program
- Waitlist Group (No Intervention): The other group will consist of participants on the wait-list. Similar to those in the intervention group, participants in the waitlist group will undergo research assessments at baseline, post-therapy, and 1 month after therapy. Subsequently, they will be included in the 4-session intervention program. No measurements will be taken after the intervention.

INTERVENTIONS:
Behavioral: The DeST-ACT Trauma-Focused Acceptance and Commitment Therapy Program — The Trauma-focused psychosocial intervention program consists of 4 sessions online therapy.
  Arms: DeST-ACT Intervention Group

SUMMARY:
The aim of this study is to develop a post-earthquake, trauma-focused Acceptance and Commitment Therapy (ACT)-based psychosocial intervention program (DeST-ACT) and to examine its effectiveness, feasibility, and acceptability of this program in enhancing life satisfaction and psychological flexibility in individuals exposed to earthquake trauma.

In this regard, the main hypothesis is that the DeST-ACT psychosocial intervention program is effective, feasible, and acceptable among individuals exposed to earthquake trauma, including both primary and secondary outcomes of the program.

DETAILED DESCRIPTION:
This quantitative, randomized controlled trial involves two groups and includes a pre-test and repeated post-tests. The study aims to assess the effectiveness, feasibility, and acceptability of the developed DeST-ACT program in addressing post-traumatic stress disorder, psychological flexibility, life satisfaction, values-based living, and depression-anxiety-stress levels in individuals affected by the February 6, 2023 earthquake. Participants will be randomly assigned to experimental and control groups in a 1:1 ratio using an internet-based block randomization program.

The DeST-ACT psychosocial intervention program consists of a 4-session online intervention supported by self-help materials. Each session in the 4-week program is held once a week for 50 minutes.

The main hypotheses are:

* The intervention group will demonstrate a significant decrease in Post Traumatic Stress Disorder (PTSD) and depression-anxiety-stress levels compared to the control group.
* The intervention group will experience a greater increase in values-based living, life satisfaction, and psychological flexibility over time compared to the control group.
* The intervention group will demonstrate a significant decrease in PTSD and depression-anxiety-stress levels compared to baseline measures.
* The intervention group will experience a greater increase in values-based living, life satisfaction, and psychological flexibility over time compared to baseline measures.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the research
* Being present in cities such as Kahramanmaras, Gaziantep, Hatay, Adiyaman, or Malatya during the earthquake on February 6, where destruction occurred
* Being literate
* Being able to have an online interview with the therapist
* Having sub-threshold PTSD or PTSD

Exclusion Criteria:

* Being in other cities at the time of the earthquake and not being exposed to the earthquake
* Having visual and/or hearing problems
* Having any psychotic disorder, experiencing an active mood episode, or having conditions such as intellectual disability or dementia that would prevent participation in therapy
* Starting a new psychiatric treatment during the research period or having a change in medication or dosage within the last 3 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
PTSD Checklist for Diagnostic and Statistical Manual of Mental Disorders-5 (PCL-5) | At baseline, after 4 weeks, after 8 weeks
  The PCL-5 was developed based on the diagnostic criteria in the Diagnostic and Statistical Manual of Mental Disorders-5, and its aim is to evaluate PTSD symptoms. The scale consists of 20 items rated on a 5-point Likert scale. Scores above 47 are indicative of PTSD.
Depression Anxiety and Stress Scale 21 (DASS-21) | At baseline, after 4 weeks, after 8 weeks
  The DASS-21 measures the dimensions of depression, stress, and anxiety. The scale consists of 21 items rated on a 4-point Likert scale ranging from 0 (Never) to 4 (Always) with scores ranging from a minimum of 0 to a maximum of 84. The Cronbach's alpha values for the scale, based on Turkish validity and reliability studies, are 0.80 for anxiety, 0.82 for depression, and 0.75 for stress.
Engaged Living Scale | At baseline, after 4 weeks, after 8 weeks
  The Engaged Living Scale is designed to evaluate values-based living. It consists of 16 items rated on a 5-point Likert scale, ranging from 1 (Totally Agree) to 5 (Totally Disagree), with scores ranging from a minimum of 16 to a maximum of 80. The scale, for which Turkish validity and reliability studies have been conducted, has two sub-dimensions: "valued living" and "life fulfillment." The Cronbach's alpha value for the Turkish version of the scale is 0.91, with 0.87 for the valued living sub-dimension and 0.86 for the life fulfillment sub-dimension.

SECONDARY OUTCOMES:
Acceptance and Action Questionnaire-2 (AAQ-2) | At baseline, after 4 weeks, after 8 weeks
  The AAQ-2 is a measure designed to evaluate experiential avoidance. The scale consists of 7 items rated on a 7-point Likert scale, with scores ranging from a minimum of 7 to a maximum of 49. Higher scores indicate greater experiential avoidance.
Therapy Satisfaction Questionnaire | after 4 week
  It is a semi-structured form designed by the researchers to assess acceptability and perceived effectiveness. The form consists of 10 questions, each scored on a scale from 0 (not at all) to 4 (completely).
Drop Rate | after 8 weeks
  To evaluate acceptability, participants' attendance rates to the program will be recorded.

OTHER OUTCOMES:
Clinician-Administered PTSD Scale for Diagnostic and Statistical Manual of Mental Disorders-5 (CAPS-5) | The scale will be used to assess the inclusion criterion before the randomization.
  Caps-5 is a structured clinical interview form developed to assess PTSD symptoms and symptom severity. The CAPS-5 consists of questions that assess the frequency and severity of each symptom, the impact of the symptoms on the patient's social and occupational functioning, and the total severity of symptoms. Turkish validity and reliability study was conducted and Cronbach's Alpha values were higher than 0.87 for all symptom dimensions.

CONTACTS AND LOCATIONS:
Locations (1):
- Cansagligi Foundation Center for Contextual Behavioral Science, Istanbul, Uskudar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No